CLINICAL TRIAL: NCT03032822
Title: Opioid Consumption After Hospital Discharge in Cystectomy Patients
Brief Title: Opioid Consumption in Cystectomy Patients
Status: Terminated | Type: Observational
Why Stopped: Unable to collect accurate opioid consumption after discharge
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Tristan Weaver, Assistant Professor - Clinical, Ohio State University
Other Study IDs: 2017H0430
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2024-03

CONDITIONS: Cystostomy; Complications; Opioid Use
Keywords: Opioid consumption; postdischarge; cystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- All Patients: All cystectomy patients who consent for the study

SUMMARY:
At the Ohio State University, and across the country, surgical patients admitted to the hospital are over-prescribed a significant amount of opioid medications upon discharge to home. Recent studies reveal that a large percentage of patients prescribed opioid medications after surgery have approximately half of the prescribed medication left over. This study aims to evaluate reported opioid use after surgery in patients undergoing cystectomy in order to better approach the issue with current opioid use and abuse trends while still providing adequate medical care and pain management to patients.

DETAILED DESCRIPTION:
Previous studies show that 67% of patients prescribed opioid medications in urologic procedures and surgeries had leftover opioid medications with a mean use of about half the medications prescribed. A similar study in thoracic surgery patients reported similar results with 71% of patients admitting to taking half or less of their prescribed opioid medications. Recent advancements in cystectomy protocol have already shown promise with reducing hospital length of stay from eight to four days, including the simultaneous reduction of opioid analgesics for pain management, with 4.9 mg morphine equivalents per day when using enhanced recovery techniques compared to 20.67 mg in traditional care. Results of the current prospective study could further support these results and include low to no risk assessments and follow-up phone calls. This study is observational and involves consenting adult patients undergoing cystectomy to pre-operative assessments including the Self Administered Gerocognitive Exam (SAGE) questionnaire, a cognitive test to identify mild-moderate cognitive impairment, and collection of demographic data and medical history. Phone call follow-ups include assessments of post-discharge pain and opioid consumption, and completing verbally an adapted Activities of Daily Living questionnaire. No additional risks have been identified by participating in this study. Participants may not directly benefit from participating in this trial, but the data collected could provide valuable insight into the discrepancy between required opioid pain medications and opioid pain medication prescription for adequate pain management. This insight could then be applied to reevaluate post-discharge pain management procedures and standards of care, therefore curbing opioid use and abuse trends

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cystectomy
* Capable and willing to consent
* Participants literate in English language

Exclusion Criteria:

* History of drug and/or alcohol abuse/dependency
* Ketamine use during hospitalization
* Illiteracy
* Presence of a clinically diagnosed major psychiatric condition such as bipolar disorder, uncontrolled major depression, schizophrenia
* Any condition that the principle investigator may disqualify the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at the OSUMC, 18 years of age and older scheduled to undergo a cystecotomy, who give written informed consent to participate in the study and who meet all inclusion and no exclusion criteria
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
opioid consumption over time | once per week, up to six weeks after surgery
  The opioid medication (oral morphine equivalent) taken by the patients will be assessed every week until the sixth postoperative week, to compare it with the amount prescribed by the physicians

CONTACTS AND LOCATIONS:
Overall Officials: Tristan E Weaver, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Efforts will be made to keep patient information confidential. individual participant data will only be available to researchers who are approved by the Institutional Review Board (IRB) to participate in study enrollment, follow up and data analysis.